CLINICAL TRIAL: NCT07395076
Title: Study of the Immunological Pathophysiological Mechanisms Associated With Acute Respiratory Distress Syndrome
Acronym: IMMUNORESP2
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP251692
Record Dates: First submitted 2026-01-09; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: acute respiratory distress syndrome; subphenotypes; ADRS
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
About 10% of patients admitted to the ICU suffer from ARDS, with a mortality rate of around 35-45%. The lack of therapeutic innovation in ARDS can be partly explained by the heterogeneity of patients included under this definition.

A better understanding of the pathophysiological mechanisms underlying the different patient phenotypes is essential to develop new therapeutic strategies.

Objectives:

To characterize the inflammatory profile of patients with ARDS using circulating biomarkers and single-cell RNA sequencing of pulmonary immune cells.

The investigators hypothesize that there is a correlation between the profile of serum biomarkers (inflammatory sub-phenotypes), the transcriptome of pulmonary immune cells.

Briefly the experimental scheme is as follow:

* Population: patients with ARDS under invasive mechanical ventilation in the ICU.
* Intervention:

  1. Determination of the inflammatory subphenotype on circulatory inflammatory biomarkers.
  2. Characterization of inflammation by single cell RNA sequencing on lung immune cells collected on broncho-alveolar fluid.

DETAILED DESCRIPTION:
Acute Respiratory Distress Syndrome (ARDS) is the most severe form of pulmonary failure. It is defined by bilateral radiologic opacities associated with severe hypoxemia, confirmed by a PaO₂/FiO₂ ratio <300 in the absence of a cardiac cause. About 10% of patients admitted to the Intensive Care Units (ICU) develop ARDS, and this diagnosis is associated with an in-hospital mortality of 35-45%. Like sepsis, ARDS leads to long-term complications. It is associated with physical deconditioning and reduced quality of life that can persist up to five years after the episode. Survivors are readmitted to the ICU within a year in 30% of cases. Moreover, excess mortality among ARDS survivors is attributable, in nearly one-third of cases, to a new acute respiratory infection.

The lack of therapeutic advances in ARDS has led researchers to better characterize patients with this condition. Different subphenotypes have been identified based on plasma inflammatory biomarker profiles, which are associated with distinct responses to treatments (such as corticosteroids, ventilatory management, and fluid management) and variable prognoses. The mechanisms underlying these different biological subphenotypes remain unknown. To further explore this concept, it is necessary to precisely identify subpopulations of patients who present with similar clinical features but distinct biological phenotypes driven by unique pathophysiological mechanisms. Establishing these different ARDS endotypes is essential for the development of innovative and targeted therapeutic strategies.

Our hypothesis is that the different biological subphenotypes of ARDS reflect distinct profiles of pulmonary immune cell populations, representing a first step toward understanding ARDS endotypes.

Identifying these endotypes is a crucial step for developing targeted and innovative therapeutic strategies aimed at reducing ARDS-related morbidity and mortality. This is the objective of the proposed project.

ELIGIBILITY:
Inclusion Criteria:

* ARDS risk factors: bacterial or viral pneumonia, extrapulmonary infection, major trauma, transfusion, inhalation injury, or shock.
* Pulmonary edema not explained by a cardiogenic cause or volume overload.
* Onset of respiratory symptoms within <7 days.
* Bilateral pulmonary involvement on chest X-ray, CT scan, or ultrasound.
* PaO₂/FiO₂ ≤ 300 assessed with PEEP ≥ 5 cmH₂O.

Exclusion Criteria:

* ARDS with intubation for more than 48 hours.
* Contraindications to bronchoscopy: effective anticoagulation, dual antiplatelet therapy, thrombocytopenia <50 G/L.
* Pre-existing immunodeficiency: active solid tumor or remission <5 years, active hematologic malignancy or remission <5 years, systemic disease (even without specific treatment), solid organ or bone marrow transplant, HIV infection with CD4 <200/mm³.
* Cardiorespiratory arrest with poor prognosis.
* Patients <18 year-old
* Patients under legal guardianship, curatorship, or deprived of liberty.
* Ongoing pregnancy.
* Patients without social security coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients in intensive care unit suffering from mechanically ventilated ARDS as defined by Matthay et al.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2029-02-05 (Estimated); Study Completion 2029-02-05 (Estimated)

PRIMARY OUTCOMES:
Single cell RNA sequencing of pulmonary immune cells | At baseline
  Single cell RNA sequencing of pulmonary immune cells collected during a bronchoalveolar lavage at inclusion.

SECONDARY OUTCOMES:
Mortality | At day 90
  Mortality rate at day 90
Mortality | 1 year
  Mortality rate at one year
Time without respiratory support | At day 28
  Number of days alive without mechanical ventilation on day 28 after inclusion or on discharge from intensive care if this occurs before the 28th day
Length of stay in intensive care | From inclusion to ICU discharge up to 1 year
  Number of days in intensive care.
Number of secondary infections | At day 90
  Rate of secondary infections defined as a new prescription of antibiotics
Number of secondary infections | 1 year
  Rate of secondary infections defined as a new prescription of antibiotics
Impact perceived on quality of life | At day 90
  Quality of life assessed though the SF-12 questionnaire on the phone.
Impact perceived on quality of life | 1 year
  Rate of secondary infections defined as a new prescription of antibiotics
Dsypnea scale | At day 90
  Dyspnea scale assessed through mMRC questionnaire on the phone
Dsypnea scale | 1 year
  Dyspnea scale assessed through mMRC questionnaire on the phone
Organ failure | At baseline
  SOFA score assessment
Organ failure | At day 7.
  SOFA score assessment
Need for vasopressor | At baseline
  Need for vasopressor (epinephrine or norepinephrine)
Vasopressor free days | At day 28 or at discharge from intensive care
  Number of days alive without vasopressors on day 28 after inclusion or on discharge from intensive care if this occurs before the 28th day.

IPD SHARING:
Plan to Share IPD: Undecided